CLINICAL TRIAL: NCT04135703
Title: Prevention of OUD: The HOME (Housing, Opportunities, Motivation and Engagement) Randomized Trial
Brief Title: Prevention of OUD: The HOME Project (Housing, Opportunities, Motivation and Engagement)
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019B0287; UH3DA050174 (NIH)
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-01

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Housing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk Prevention Services +Housing (Experimental): Opioid and related prevention services including Strengths-Based Outreach and Advocacy (SBOA), MI, HIV risk and suicide prevention (CTSP) as well as rental and utility assistance for 6 months.
  Interventions: Behavioral: Risk Prevention Services + Housing
- Risk Prevention Services Only (Experimental): Opioid and related prevention services including Strengths-Based Outreach and Advocacy (SBOA), MI, HIV risk and suicide prevention (CTSP).
  Interventions: Behavioral: Risk Prevention Services Only

INTERVENTIONS:
Behavioral: Risk Prevention Services + Housing — opioid and related prevention services in addition to 6 months of rental assistance
  Arms: Risk Prevention Services +Housing
Behavioral: Risk Prevention Services Only — opioid and related prevention services for 6 months
  Arms: Risk Prevention Services Only

SUMMARY:
Homeless youth have a much higher rate of substance use than non-homeless peers with evidence suggesting that homeless youth have the highest rates of opioid use among youth subgroups in the country (Brands et al., 2005); heroin using homeless youth also appear to have the highest rates of IV drug use and HIV (Rhoades et al., 2014). Given the high rates of opioid use, exposure to violence, mental and physical health challenges, and high rates of mortality in homeless youth, it is surprising that no study to date utilizes a randomized controlled design to test prevention of opioid and other drug use among this vulnerable population. Resolution of youth homelessness through housing and prevention services, often referred to as "Housing First", as proposed in the current study, has great potential to reduce the likelihood for the development of an opioid use disorder as well as other problem behaviors associated with living on the streets. However, only 20-30% of homeless youth samples report ever having stayed at a crisis shelter, 9% report having ever accessed mental health services, and 15% report ever having received substance use treatment (Ray, 2006) indicating a need to reach and engage youth in services that are feasible and acceptable. This study will provide essential information for researchers and providers on the efficacy of housing + opioid and related risk prevention services in an RCT on opioid use, how moderators affect the response, and mechanisms underlying change.

DETAILED DESCRIPTION:
The overarching goal of this application is to evaluate a comprehensive intervention for the prevention of opioid use disorder and for increasing other resilient outcomes in this special population of high-risk young adults. Phase I of the study includes a nonrandomized pilot study with a sample of 21 youth to assess initial efficacy, feasibility of recruitment and acceptability of the housing + opioid and related risk prevention services. Upon meeting transition milestones, 240 youth will be randomized into housing + opioid and related risk prevention services versus opioid and related risk prevention services alone for Phase II. In this study, we seek to determine if adding housing to opioid and related risk prevention services yields a significant benefit above and beyond the benefit yielded by opioid and related risk prevention services alone. Phase II follow-up will be conducted at 3, 6, 9 and 12-months post-baseline to assess stability of effects. Sample inclusion criteria, recruitment and screening will be identical for both phases, as described below. The unique components of Phase I and Phase II are then described separately.

Sample Inclusion Criteria.

1. We will include youth between the ages of 18 to 24 years.
2. Youth meets the criteria for homelessness as defined by the federal McKinney-Vento Act (2002) as "lacking a fixed, regular, stable, and adequate nighttime residence" and includes "living in a publicly or privately operated shelter designed to provide temporary living accommodations, or a public or private place not designed for, or ordinarily used as, regular sleeping accommodations for human beings."
3. Youth fails to meet DSM 5 criteria for Opioid Use Disorder as assessed by the SCID (First et al., 2015).
4. Those who report suicide ideation on the Scale for Suicide Ideation - Worst Point (SSI-W) (Beck, Brown, & Steer, 1997) will also receive suicide prevention.

Participant recruitment and sample availability. Service-connected youth will be recruited from the drop-in and adult shelters, non-service connected youth will be recruited through outreach to local soup kitchens, sandwich lines, the streets, parks and library. Given the high rates of homeless youth in Columbus, we do not anticipate any recruitment problems.

Screening and intake. Project staff will maintain offices within the drop-in center. Youth who are engaged on the streets will be transported to the drop-in center. An RA will engage and screen youth to determine basic eligibility for the study. After the brief screening and stated interest in the project, written consent will be obtained and the Structured Clinical Interview for DSM-5 Disorders (SCID) (First, Williams, Karg, & Spitzer, 2015) section on Opioid Use Disorder, will be administered to determine formal eligibility.

The Community Advisory Group, including homeless providers, homeless youth, landlords, substance use treatment experts and policy makers will meet throughout the project period, shaping study procedures, and easing transition of intervention to practice by the end of the study.

Phase I (UG3) Using the same recruitment strategy, eligibility criteria and assessment package (including stress biomarkers) as Phase II, a non-randomized pilot of the housing + opioid and related risk prevention services intervention (N = 21) will be completed in year 1. The sample size of 21 reflects three months of recruitment of seven youth/month. All youth will receive the 6-month housing + opioid and related prevention services intervention. Youth will be assessed at baseline, 3 and 6-months using the proposed assessment battery, and qualitative interviews. The primary purpose of this phase is to document feasibility of recruitment, acceptability of the intervention, and initial pre-post change on targeted outcome measures. As the housing + prevention services and assessment battery are identical in Phase 1 and Phase II, they are described in detail following the description of Phase II. Those aspects unique to Phase I are discussed immediately below.

Phase I: Assessment of acceptability, feasibility and initial efficacy of the intervention. Acceptability of the intervention will be assessed by the retention of youths in the intervention, the total number of advocacy sessions attended, length of time remaining in project supported housing, and by the percentage of eligible youth who agree to participate in the study. In addition, the extent to which landlords consent to continuing participation in the second phase of the trial is essential. Assessment of feasibility includes documentation of 1) whether participants can be recruited, engaged, and maintained in the housing + opioid and related risk prevention services as proposed, data which can be obtained from RA screening forms and advocate records (meetings attended, maintenance of housing), and 2) whether the timeline proposed for housing youths (anticipated to average 4 weeks, and time to housing will be tracked) and other intervention procedures can be maintained as proposed. In order to estimate initial efficacy, we will assess youth at baseline, 3 and 6-months to determine change in identified targeted outcomes (e.g. opioid and other substance use, homelessness and related problems). In addition to the quantitative analysis, qualitative interviews with each youth will provide a fuller understanding of the youths' response to the intervention.

Phase I: Quantitative Analysis. Repeated measures ANOVA will be used to test the efficacy of the intervention (time effects). Three testing occasions (e.g., baseline, 3, and 6 months) will be the within-subject dependent variables. The primary outcome is opioid use, and secondary outcomes are listed below under "dependent variables." It is predicted that there will be a main effect of time; youth will show reductions in opioid use, and improved functioning in other domains at post-intervention (6-months).

Phase I: Qualitative Analysis. In order to increase our understanding of youths' response to the intervention such as experiences associated with differing levels of housing success and satisfaction with services, each youth at 6 months post-baseline will be interviewed regarding their experiences in the study. Supplementing the quantitative findings, interviews can provide better understanding of factors that promote engagement and success among youth as well as factors that prevented youth from successfully maintaining their housing. Additionally, qualitative data can help explain any unexpected findings, and provide a greater richness when reporting and interpreting the quantitative outcomes.

Phase II (UH3) In Phase II, 240 homeless youths between the ages of 18 to 24 years recruited from the streets and drop-in center will be randomly assigned to 1) 6-months of housing + opioid and related risk prevention services (n = 120), or to 2) opioid and related risk prevention services alone (n = 120). In addition, all youth will be screened using the Scale for Suicide Ideation - Worst Point (SSI-W). We expect that approximately N =100 youth will report suicidal ideation and those youth will also receive the suicide prevention intervention.

Using an intent to treat design, follow-up assessments will be completed at 3, 6, 9 and 12 months post-baseline. Four advocates will provide services so that advocate effects can be examined (Baldwin et al., 2011), and each advocate will provide all opioid and related risk prevention services to the youth on their caseload. Advocates will be crossed by condition to "equate" conditions on advocate characteristics. RA's will be blind to condition at all assessment timepoints.

Project Intervention: Housing + Prevention Services versus Prevention Services alone Housing + Opioid and Related Risk Prevention Services integrates independent housing, Strengths-Based Outreach and Advocacy (SBOA), HIV prevention and MI (Miller & Rollnick, 2012) and Cognitive Therapy for Suicide Prevention (CTSP). Each component of the intervention is described below.

Strengths-Based Outreach and Advocacy (SBOA). SBOA focuses on identifying and engaging youth from the streets and drop-ins/shelters etc. and assisting these youth to meet their basic needs (i.e., referrals to food pantries), obtain government entitlements (i.e., SSDI/SSI, cash assistance, food stamps), and connect to other needed supports (education, job training). The advocates provide referrals and/or transport youth to appointments as needed. The initial meeting provides an opportunity to gather information. The advocate will review each of six general areas with the youth to gather a history and picture of the current situation: (1) housing needs; (2) health care; (3) food; (4) legal issues, (5) employment and (6) education. The advocate will assist youth assigned to the opioid and related risk prevention services only comparison condition to obtain housing within the community, as is usually provided with SBOA, but unlike the youth in the housing intervention, they are not provided housing by the project. Once this review is complete, an initial intervention plan is developed with specific goals and objectives. Advocates are available 24 hours for crises.

HIV prevention. Every youth will receive the 2-session intervention which uses cognitive-behavioral techniques with a focus on skills building/behaviors (role plays with condom application, cleaning needles, communication/negotiation and problem solving), used in prior projects with homeless youth with success reducing risk behaviors (e.g., Carmona et al., 2014; Slesnick & Kang, 2008).

Motivational Interviewing (MI). The Project Match manual was adapted for homeless/runaway youth in prior trials in consultation with William R. Miller and Bo Miller (NIAAA grant no. R01AA12173 and NIDA grant R29DA11590). Adaptation of the manual included attention to the unique life situation of homeless youth in understanding motivations and challenges to recovery while homeless. Session 1 begins with a period of open-ended MI, to establish therapeutic rapport and elicit client change talk. In session 2 the advocate continues to focus on enhancing intrinsic motivation for change, developing discrepancy, transitioning as appropriate into the negotiation of a change plan and evoking commitment to the plan.

Cognitive Therapy for Suicide Prevention (CTSP). The Cognitive Therapy Intervention for Suicide Attempters, developed by Aaron Beck, Gregory Brown and Amy Wenzel (Wenzel, Brown, & Beck, 2009) has shown promising results for both adults (Brown et al., 2005) and youth (Brent et al., 1993; Stanley et al., 2009). This approach is innovative in that suicidal behavior is the primary target for treatment, rather than being secondary to an underlying psychological disorder, which has been the standard in the field (Wenzel et al., 2009). As a short term treatment (10 sessions), the intervention is particularly feasible for youth who have high rates of treatment refusal and drop-out. CTSP is based upon the theoretical assumption that the manner by which people think and interpret their life events determines their emotional and behavioral responses to those events. Hence, maladaptive cognitions associated with suicidal ideation are the primary focus of the treatment.

Housing. Those randomized to receive housing + opioid and related risk prevention services will receive each prevention component above, plus 6-months of housing. The advocate will work with the youth to identify appropriate housing among the available choices. The project will cover damage deposit, application fees (including FABCO report, credit report), and will automatically pay the landlords the rental checks at the beginning of each month. As in the prior Stage 1 and 2 studies, Nationwide Children's Hospital will not sign leases on behalf of the youth, and so the youth will sign the lease.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18 to 24 years
* meets McKinney-Vento definition of homeless
* fails to meet DSM 5 criteria for Opioid Use Disorder as assessed by the SCID

Exclusion Criteria:

-

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] Ahrens K, Blackburn N, Aalsma M, Haggerty K, Kelleher K, Knight DK, Joseph E, Mulford C, Ryle T, Tolou-Shams M. Prevention of Opioid Use and Disorder Among Youth Involved in the Legal System: Innovation and Implementation of Four Studies Funded by the NIDA HEAL Initiative. Prev Sci. 2023 Oct;24(Suppl 1):99-110. doi: 10.1007/s11121-023-01566-6. Epub 2023 Jul 1. PMID 37393415
- [Derived] Chavez L, Kelleher K, Bunger A, Brackenoff B, Famelia R, Ford J, Feng X, Mallory A, Martin J, Sheftall A, Walsh L, Yilmazer T, Slesnick N. Housing First Combined with Suicide Treatment Education and Prevention (HOME + STEP): study protocol for a randomized controlled trial. BMC Public Health. 2021 Jun 12;21(1):1128. doi: 10.1186/s12889-021-11133-9. PMID 34118916
- [Derived] Slesnick N, Chavez L, Bunger A, Famelia R, Ford J, Feng X, Higgins S, Holowacz E, Jaderlund S, Luthy E, Mallory A, Martin J, Walsh L, Yilmazer T, Kelleher K. Housing, opportunities, motivation and engagement (HOME) for homeless youth at-risk for opioid use disorder: study protocol for a randomized controlled trial. Addict Sci Clin Pract. 2021 May 12;16(1):30. doi: 10.1186/s13722-021-00237-7. PMID 33980315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 394 youth approached, 240 eligible and enrolled.
Pre-assignment Details: Failed: (n=154)
  * Not homeless (n=20)
  * Over the age of 24 (n=2)
  * Under the age of 18 (n=7)
  * Met DSM 5 criteria for OUD (n=27)
  * Declined Participation (n=39)
  * Failed to return (n=43)
  * Refused to wear a mask during intake (n=1)
  * Unable to focus to complete intake (n=1)
  * Difficulty/unable to answer questions (n=5)
  * Could not show proof of Guardianship (n=2)
  * Had difficulty understanding the project/process (n=7)
Groups:
- Risk Prevention Services +Housing: Opioid and related prevention services included Strengths-Based Outreach and Advocacy (SBOA), MI, HIV risk and suicide prevention (CTSP) as well as rental and utility assistance for 6 months.
- Risk Prevention Services Only: Opioid and related prevention services included Strengths-Based Outreach and Advocacy (SBOA), MI, HIV risk and suicide prevention (CTSP).
Period: Overall Study
Arm/Group | Risk Prevention Services +Housing | Risk Prevention Services Only
Started | 120 | 120
Completed | 120 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recruited as proposed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risk Prevention Services +Housing | Risk Prevention Services Only | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant age measured continuously
  years | 21.8 (1.84) | 20.93 (1.82) | 21.05 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth, categorical
  Participants
    Female | 64 | 53 | 117
    Male | 56 | 67 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (NIH/OMB) self-report
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 5 | 2 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 65 | 72 | 137
    White | 25 | 30 | 55
    More than one race | 21 | 15 | 36
    Unknown or Not Reported | 2 | 1 | 3
% days opioid use in prior 90 days [Mean (Standard Deviation); unit: % of days of opioid use in prior 90 days] — Percent of days opioid use measured using the Form 90
  % of days of opioid use in prior 90 days | .35 (.30) | .32 (.25) | .335 (.275)

OUTCOME MEASURES:

1. Primary Outcome: Frequency (% Days) of Opioid Use in Prior 3 Months
Description: frequency (% days in prior 90) of opioid use is measured at baseline, 3, 6, 9 and 12 months post-baseline
Time Frame: 12 months
Population: Frequency of opioid use in prior 90 days (percentage of days use) was assessed at each follow-up point (3, 6, 9 and 12-months post-baseline) using the Form 90 interview.
Measure: Mean (Standard Deviation); unit: % days opioid use
Arm/Group | Risk Prevention Services +Housing | Risk Prevention Services Only
Number analyzed (Participants) | 120 | 120
% days opioid use | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: From enrollment to 12-month follow-up.
Arm/Group | Risk Prevention Services +Housing | Risk Prevention Services Only
All-Cause Mortality (participants affected / at risk) | 4/120 | 1/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT04135703/Prot_SAP_000.pdf